CLINICAL TRIAL: NCT02645942
Title: L-carnitine for Reducing Cardio-metabolic Risk in Patients With Obstructive Sleep Apnea - Double Blind Randomized Clinical Trial
Brief Title: L-carnitine for Reducing Cardio-metabolic Risk in Patients With Obstructive Sleep Apnea
Acronym: CARNIMET
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to organization reasons.
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pawel Bogdanski, Ass. Prof, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 962/15
Record Dates: First submitted 2015-12-29; First posted 2016-01-05 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Carnitine; placebo; risk factors
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): L-carnitine 1400 mg daily for 8 weeks
  Interventions: Dietary Supplement: L-carnitine
- Placebo group (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-carnitine — L-carnitine 1400 mg daily for 8 weeks
  Arms: Intervention group
Dietary Supplement: Placebo — Placebo daily for 8 weeks
  Arms: Placebo group

SUMMARY:
The investigators designed this intervention to investigate the potential role of L-C in lipid and carbohydrates metabolism (primary outcome) with precision noninvasively measurement of: central blood pressure, pulse wave velocity and peripheral arterial stiffness (secondary outcome) in OSA patients.

DETAILED DESCRIPTION:
After screening all patients will be randomized in 1:1 ratio to either placebo group or study group (receiving L-C for 8-weeks). Randomization will stratify patients by: age, sex, BMI and severity of OSA. Randomized patients will receive orally either placebo or L-C once a day for 8-weeks. All supplements will be packed in a white box. Because this is a double-blind study, vial labels will contain a unique identification number that will not disclose to the patient or investigator if L-C or matching placebo is included. The daily amount of L-C will be 1400 mg. The detailed composition of the product will be assessed. All patients will receive a test product during the control visits once a month and will be asked to take it once a day in the morning. The completion of the data will be checked during the visits and also via telephone while the study is conducted. All concomitant medications used (including herbal supplements) will be recorded in electronic database. The patients will be asked to continue their habitual diet. Moreover, they will be also advised that they are free to withdraw from participation in this study at any time, for any reason, and without prejudice. The reason for withdrawal and the date of discontinuation will be recorded in our database. Any Adverse Event (AE) will be recorded according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE), clinically significant AE, severe laboratory abnormality, intercurrent illness, or other medical condition that indicates that continued administration of study medication is not in the best interest of the patient.

The treatment will be administrated under supervision of experienced nutritionist and medical doctor. The anthropometrical and biochemical measurements with assessment of diet, quality of life and sleep will be completed by the patients at each of the study visits, which will take place at the baseline (screening visit), after 4 weeks, in the post-intervention period (week 8) and at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed OSA classified according to the apnea hypopnea index (AHI) as a mild (5.0-14.9), moderate (15.0-29.9), and severe (≥30.0 events per hour),
* treatment with Continuous Positive Airway Pressure (CPAP) for at least 6 months before study screening,
* disturbed lipid metabolism (according to the National Health and Nutrition Examination Survey: LDL-C>100 mg/dl, or TG>150 mg/dl) or use of hypolipidemic drugs,
* disturbed glucose metabolism (Diabetes mellitus or impaired glucose tolerance or impaired fasting glucose) according to American Diabetes Federation or use of hypoglycaemic drugs,
* willingness to participate in the study,
* age over 18,
* continued habitual diet during the study period,
* performance status ≥ 80 according to Karnofsky score

Exclusion Criteria:

* newly diagnosed OSA and individuals treated with CPAP,
* other than OSA lung dysfunctions,
* do not use of hypoglycaemic and hypolipidemic drugs,
* modification of hypolipidemic or hypoglycaemic treatment during the study period,
* pregnancy or lactation,
* cancer (excluding curatively treated with no evidence of diseases for 5 years),
* severe liver and kidney diseases (Aspartate aminotransferase (ASPAT) and alanine aminotransferase (ALAT) >3 × the upper limit of normal (ULN), Bilirubin >1.5 × ULN, Creatinine >1.5 × ULN),
* known sensitivity to any component of the product,
* diagnosed CVD (myocardial infarct, stroke, angina pectoris).
* an active drug or alcohol abuse,
* legal incompetence,
* limited legal incompetence,
* any uncontrolled medical condition that may put studied patients at high risk during study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Changes in Total cholesterol, LDL cholesterol, HDL cholesterol and Triglycerides concentration | 6 months
Changes in fasting glucose concentration | 6 months
Changes in insulin concentration | 6 months

SECONDARY OUTCOMES:
Changes in central blood pressure | 6 months
Changes in pulse wave velocity | 6 months
Changes in peripheral arterial stiffness | 6 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Bogdański, Ass Prof, MD, Principal Investigator — Poznan University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No